CLINICAL TRIAL: NCT02603796
Title: 3D Imaging of Neonatal Subjects
Brief Title: 3D Imaging of Neonatal Faces
Status: Completed | Type: Observational
Sponsor: Sharp HealthCare (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Principal Investigator, Anup Katheria, M.D., Director of Neonatal Research, Sharp HealthCare
Other Study IDs: 3D Imaging in neonates
Record Dates: First submitted 2015-10-30; First posted 2015-11-13 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Nose Deformities, Acquired
Keywords: 3-Dimensional; continuous positive airway pressure; nasal changes
MeSH Terms: conditions — Nose Deformities, Acquired

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Newborns requiring ncpap: 3D scan of nares will be performed before and after administration of NCPAP for infants with Corrected Gestational Age greater than or equal to 24 weeks and less than or equal to 42 weeks.
  Interventions: Other: 3D Scan of nares

INTERVENTIONS:
Other: 3D Scan of nares — 3D scan of subjects nose prior to implementation of ncpap and upon discontinuation of ncpap.

SUMMARY:
Facial scans of newborns will be performed before and after implementation of respiratory support devices such as nasal CPAP. 3D scanned images will be processed by Fisher & Paykel Healthcare Limited. Images will be analyzed for changes or distortion in nasal structure.

DETAILED DESCRIPTION:
Any newborns admitted to the neonatal intensive care unit at Sharp Mary Birch Hospital for Women and Newborns between 24-42 weeks CGA with parental informed consent are eligible. 3D scanned image will be obtained prior to implementation of nasal support devices and after nasal support devices. Fisher & Paykel Healthcare Limited will analyze the 3D images and observations will be made for changes in nasal structure or distortion.

ELIGIBILITY:
Inclusion Criteria:

* Infants between 24 and 42 weeks corrected gestational age (inclusive) born at Sharp Mary Birch NICU,
* Signed informed consent form

Exclusion Criteria:

* Nasally intubated infants
* Infants with craniofacial abnormalities

Ages: 24 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants between 24 and 42 weeks corrected gestational age and admitted to Sharp Mary Birch NICU.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2015-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Deformation changes in nares of preterm infants that require ncpap | Up to 6 months
  3D scans of infants face will be performed before implementation of NCPAP and a 3D scan will be performed after the NCPAP is discontinued and the images will be analyzed for changes in facial structures that might be due to NCPAP.

OTHER OUTCOMES:
Gestational Age at time of CPAP | Up to 6 months
Photograph of nose with scaled ruler | Up to 6 months
Initial 3D scan | Up to 6 months
  Date & time of scan, head circumference, CGA, current weight, nasal integrity
Post ncpap 3D scan | Up to 6 months
  Date & time of scan, head circumference, CGA, current weight, nasal integrity and/ or any notable distortion
Total duration of ncpap days | Up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sharp Mary Birch Hospital for Women and Newborns, San Diego, California, United States